CLINICAL TRIAL: NCT06699537
Title: Effectiveness of Lacticaseibacillus Rhamnosus LRa05 in Alleviating Allergic Rhinitis and Its Impact on Gut Microbiota: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Lacticaseibacillus Rhamnosus LRa05 for Alleviating Allergic Rhinitis in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK2024016
Record Dates: First submitted 2024-11-15; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Allergic Rhinitis (AR)
MeSH Terms: conditions — Rhinitis, Allergic | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double(Participant,Investigator)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Participants in the probiotic group received 1 sachet probiotic product per day.
  Interventions: Dietary Supplement: probiotic product
- Placebo group (Placebo Comparator): Participants in the placebo group received 3g of maltodextrin per day.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: probiotic product — During the study, subjects take one sachet of Lactobacillus rhamnosus LRa05 daily. Evaluation is conducted by monitoring the subjects' nasal symptoms and gut microbiota before and after the intervention.
  Arms: Probiotic group
Dietary Supplement: Maltodextrin — During the study, subjects in the control group take one sachet of maltodextrin daily with 3.0g. Evaluation is conducted by monitoring the subjects' nasal symptoms and gut microbiota before and after the 8-week trial.
  Arms: Placebo group

SUMMARY:
The clinical trial aims to investigate the efficacy of Lactobacillus rhamnosus LRa05 in alleviating allergic rhinitis and its impact on the gut microbiota among 70 pediatric participants aged 4-12. The primary objective is to validate the improvement in allergic rhinitis symptoms following an 8-week intervention with Lactobacillus rhamnosus LRa05. Participants were instructed to consume the probiotic powder daily for approximately 8 weeks. At baseline, week 4, and week 8 endpoints, assessments of nasal symptoms, quality of life questionnaires, and stool samples for microbiota analysis were conducted on the participants, and blood samples were collected for immune-related factor testing.

DETAILED DESCRIPTION:
Research has indicated that allergic rhinitis (AR) is associated with a decrease in the diversity of the gut microbiota, particularly in children, potentially linking to the development of allergic diseases. Preclinical studies have shown that supplementation with Lactobacillus rhamnosus LRa05 can regulate immune responses, inhibit inflammatory factors, and the predictive functions of the gut microbiota suggest an increase in gene abundance within pathways related to immune modulation, anti-inflammatory effects, and maintenance of gut barrier integrity. To ascertain the effectiveness of the probiotic strain LRa05, a randomized, double-blind, placebo-controlled trial was conducted by the investigators to evaluate and gather data on alterations in the gut microbiota and allergic rhinitis symptoms among pediatric participants. The trial spanned over 8 weeks, with washout periods incorporated at the commencement and conclusion. Throughout the study, participants ingested Lactobacillus rhamnosus LRa05 and were subjected to a series of health examinations and assessments, including nasal symptom scores, quality of life questionnaires, and stool sample collections for microbiota analysis, as well as blood samples for immune-related factor testing. The primary objective was to validate the improvement in allergic rhinitis symptoms and the modulation of the gut microbiota following the intervention with LRa05.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily, in writing, sign the informed consent form, agreeing to participate in this study;
2. Capable of completing the study according to the test protocol requirements;
3. Age between 4 to 12 years old;
4. Meet the diagnostic criteria for allergic rhinitis established in the "Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (Revised Edition 2022)";
5. Symptoms: Presence of two or more symptoms such as sneezing, watery rhinorrhea, nasal itching, and nasal congestion, with symptoms lasting or accumulating for more than one hour per day, possibly accompanied by eye itching, tearing, and redness, and other ocular symptoms;
6. Signs: Nasal mucosa is pale and edematous, possibly with watery secretions;
7. Laboratory tests: At least one allergen detected by skin prick test and/or specific IgE positivity in serum;
8. No use of antihistamines, corticosteroids, or immunosuppressants in the month before screening;
9. No history of heart, liver, kidney, nervous system, mental disorders, or metabolic abnormalities.

Exclusion Criteria:

1. Use of medications affecting the gut microbiota (including antimicrobial drugs, probiotics, intestinal mucosal protective agents, traditional Chinese patent medicines, etc.) for more than 1 week within 1 month prior to screening;
2. Patients with coexisting pulmonary tuberculosis;
3. Those with coexisting allergic asthma;
4. Individuals with nasal polyps or severe nasal septal deviation;
5. Patients with severe systemic diseases or malignant tumors;
6. Those with congenital genetic diseases or congenital immunodeficiency diseases;
7. Regular use of probiotics or prebiotics within 6 months prior to the screening period;
8. Individuals with severe gastrointestinal diseases (including severe diarrhea, inflammatory bowel diseases, etc.);
9. Those with metabolic syndrome (including obesity, dyslipidemia, hypertension, diabetes, etc.);
10. Individuals with sinusitis, otitis media, or respiratory tract infections;
11. Those allergic to any components of the probiotics used in this trial;
12. Women who are pregnant or breastfeeding, or those planning to conceive in the near future;
13. Subjects who discontinue the test sample or add other medications midway, making it impossible to determine efficacy or with incomplete information;
14. Those who have recently consumed items similar to the test product, affecting the judgment of the results;
15. Subjects who, due to their own reasons, cannot participate in the trial;
16. Any other subjects deemed unsuitable to participate by the investigators.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total Nasal Symptom Score (TNSS) | 8 weeks
  The Total Nasal Symptom Score (TNSS) will be used to assess the severity of nasal symptoms in subjects. TNSS includes four symptoms: sneezing, rhinorrhea, nasal itching, and nasal congestion, each rated by the patient on a severity scale (0 points indicate no symptoms; 1 point indicates mild symptoms, easily tolerable; 2 points indicate moderate symptoms, annoying but tolerable; 3 points indicate severe symptoms, intolerable, affecting daily life and sleep). The total score is the sum of the individual symptom scores, ranging from 0 to 12, with higher scores indicating more severe symptoms. The TNSS scores at baseline and after the 8-week intervention will be recorded and the change will be calculated.
Change in Visual Analogue Scale (VAS) for Nasal Symptoms | 8 weeks
  The Visual Analogue Scale (VAS) will be used to evaluate the treatment effect in subjects. VAS scores pertain to four nasal symptoms: sneezing, rhinorrhea, nasal itching, and nasal congestion, with patients marking a point on a 0-10 cm line (0 indicates no symptoms, 10 indicates the most severe symptoms). The total score is the sum of the individual symptom scores, ranging from 0 to 40, with higher scores indicating more severe symptoms. The VAS scores at baseline and after the 8-week intervention will be recorded and the change will be calculated.
Change in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) | 8 weeks
  The Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) will be used to assess the quality of life in subjects. The RQLQ consists of 28 questions that evaluate the degree to which subjects have been bothered by problems in the past 7 days (0 points indicate not bothered at all; 1 point indicates hardly bothered; 2 points indicate occasionally bothered; 3 points indicate moderately bothered; 4 points indicate quite a bit bothered; 5 points indicate very bothered; 6 points indicate extremely bothered). The total score is the sum of the individual question scores, ranging from 0 to 168, with higher scores indicating a greater impact on quality of life. The RQLQ scores at baseline and after the 8-week intervention will be recorded and the change will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shangdong University, Jinan, Shangdong, China

IPD SHARING:
Plan to Share IPD: No